CLINICAL TRIAL: NCT00313131
Title: A Randomised Controlled Trial of Single Dose Tinidazole+Fluconazole Versus Longer Courses of Metronidazole+Clotrimazole in the Management of West African Women With Vaginal Discharge
Brief Title: Study of the Management of Vaginal Discharge in West African Using Single Dose Treatments
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Canadian International Development Agency (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUS 03-32
Record Dates: First submitted 2006-04-07; First posted 2006-04-11 (Estimated); Last update posted 2006-04-11 (Estimated); Status verified 2005-09

CONDITIONS: Bacterial Vaginosis; Candidiasis; Vaginitis
Keywords: bacterial vaginosis; vaginal candidiasis; trichomoniasis; vaginitis; Ghana; Togo; Mali; Guinea
MeSH Terms: conditions — Vaginosis, Bacterial; Candidiasis; Vaginitis; Candidiasis, Vulvovaginal; Trichomonas Infections

INTERVENTIONS:
Drug: tinidazole+fluconazole vs metronidazole+clotrimazole

SUMMARY:
This randomised controlled trial aimed to verify whether directly observed single dose treatment (with tinidazole+fluconazole) would be as effective as the longer standard treatments (metronidazole for 7 days, plus vaginal clotrimazole for 3 days) in the syndromic management of women presenting with vaginal discharge in primary health care centers of Ghana, Togo, Guinea and Mali. It was designed as an effectiveness trial, i.e. it was done under conditions typical of routine work in these health centers

DETAILED DESCRIPTION:
Abstract Objective: Evaluate whether single-dose treatments are as effective as standard therapy in the syndromic management of vaginal discharge.

Methods: A randomized controlled effectiveness trial comparing single-dose tinidazole plus fluconazole (TF) to seven days of metronidazole plus three days of vaginal clotrimazole (MC) among 1570 women presenting with vaginal discharge in primary health care institutions of Ghana, Togo, Guinea and Mali. Participants were randomly allocated to one of the two treatments by research nurses or physicians using pre-coded envelopes. Effectiveness was assessed by symptomatic response on day 14.

Findings: The two treatment regimens had similar effectiveness: complete resolution was seen in 66% (TF) and 64% (MC) and partial resolution in 33% (TF) and 34% (MC) of participants (p=0.26). Effectiveness was similar among subgroups with vulvovaginal candidiasis, T. vaginalis vaginitis or bacterial vaginosis. The two treatment regimens had a similar effectiveness among HIV-infected (TF: n=76, 71% complete resolution, 28% partial; MC: n=83, 72% complete, 25% partial, p=0.76) and HIV-uninfected women (TF: n=517, 68% complete, 32% partial; MC: n=466, 65% complete, 33% partial, p=0.20). Cervical infections with N. gonorrhoeae, C. trachomatis and M. genitalium were uncommon among women not involved in sex work, were associated with bacterial vaginosis or T. vaginalis vaginitis, and did not alter response to treatment with agents active against vaginal infections. Four fifths of women not relieved by single-dose TF had a favourable response when MC was administered as second-line treatment.

Conclusion: Single-dose TF is as effective as multiple-dose MC in the syndromic management of vaginal discharge, even among the HIV-infected. Given its low price and easier compliance, tinidazole/fluconazole should be considered as a first-line treatment of the vaginal discharge syndrome.

ELIGIBILITY:
Inclusion Criteria:

* women consulting for vaginal discharge
* local resident
* willingness and ability to consent

Exclusion Criteria:

* sex worker consulting for active screening
* main complaint of lower abdominal pain
* allergy to one of the study drugs

Min Age: 11 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1524
Dates: Start 2004-01; Study Completion 2005-05

PRIMARY OUTCOMES:
Symptomatic resolution of the vaginal discharge according to the patient

SECONDARY OUTCOMES:
Objective resolution of the vaginal discharge according to the study nurse or medical officer

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Pepin, MD, Principal Investigator — U of Sherbrooke
Locations (7):
- Ghana (2):
  - Adabraka Polyclinic, Accra
  - Suntreso Polyclinc, Kumasi
- Guinea (2):
  - Centre de Santé Carrière, Conakry
  - Centre de Santé Madina, Conakry
- Togo (3):
  - Centre de Santé d'Adakpamé, Adakpamé
  - Clinique IST d'Agoe Nyivé, Lomé
  - Clinique IST d'Amoutivé, Lomé

REFERENCES:
- [Derived] Pepin J, Sobela F, Khonde N, Agyarko-Poku T, Diakite S, Deslandes S, Labbe AC, Sylla M, Asamoah-Adu C, Frost E. The syndromic management of vaginal discharge using single-dose treatments: a randomized controlled trial in West Africa. Bull World Health Organ. 2006 Sep;84(9):729-38. doi: 10.2471/blt.06.029819. PMID 17128343